CLINICAL TRIAL: NCT02817984
Title: A Phase I Open-label Study Evaluating the Safety of Acellular Adipose Tissue (AAT), a Novel Soft Tissue Reconstruction Solution, in Healthy Volunteers
Brief Title: Safety Study of Acellular Adipose Tissue for Soft Tissue Reconstruction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00027657; CF-11 (Other Grant/Funding Number: U.S. Army Medical Research and Materiel Command); 16520 (Other: Food and Drug Administration)
Record Dates: First submitted 2016-06-21; First posted 2016-06-29 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Healthy Volunteers
Keywords: Abdominoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Group (Experimental): Participants (n=10) will be enrolled and assigned chronologically to one of five excision time points: Weeks 2 (n=10), 4 (n=2), 6 (n=2), 8 (n=2), and 12 (n=2) post-injection. Implants will be injected on Day 0. All participants will be administered up to five (5) 2 milliliter (mL) subcutaneous injections of acellular adipose tissue (AAT) via sterile injection into the area identified for planned excision. Total injected AAT volume per patient will not exceed 10 mL.
  Interventions: Biological: Acellular Adipose Tissue (AAT)

INTERVENTIONS:
Biological: Acellular Adipose Tissue (AAT) — The components of the adipose-derived scaffold are all naturally occurring AAT proteins and proteoglycans that provide a natural scaffold. The nature of the AAT also enhances host tissue integration since matrix components can be easily degraded by cell-secreted enzymes as tissue remodeling takes place. Mechanisms for matrix turnover are already established in host cells, avoiding any concerns over proper clearance of scaffold materials from the body.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of acellular adipose tissue (AAT), intended for the repair of soft tissue defects in humans, in healthy volunteers. The investigators hypothesize that AAT will be safe and well tolerated upon injection into human soft tissue.

DETAILED DESCRIPTION:
This is a 12-week, prospective, Phase I study in healthy volunteers assessing the safety and tolerability of acellular adipose tissue (AAT) intended for the repair of soft tissue defects in humans. Up to five (5) 2 milliliters (mL) subcutaneous injections of AAT will be administered into redundant tissues previously identified and scheduled for surgical removal in an elective surgical procedure.

Participants will be enrolled and assigned chronologically to one of five excision time points: Weeks 2, 4, 6, 8, and 12 post-injection. Implants will be injected on Day 0. A safety visit will occur at 1 week post-injection; follow-up visits will occur at Weeks 2 and 4 (for patients who still have implants) post-injection and at time of tissue excision. At the end of their assigned study time point, participants will have all AAT implants removed simultaneously during their elective surgery. Implants will be assessed using histopathological analyses including hematoxylin and eosin staining and flow cytometry. The primary outcome of safety will be determined by the incidence and rate of adverse / unanticipated events. Secondary outcomes include histopathological assessment of the explanted implants and tolerability determined by participant-reported comfort and physician-reported ease-of-use with the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-65 years who have sought elective surgery for the removal of redundant tissue of the abdomen (abdominoplasty or panniculectomy) or arm (brachioplasty).
* Willingness to delay elective surgery up to 12 weeks in order to participate in the study.
* Consent to photography for research purposes.
* Willingness to follow study requirements.
* Ability to give informed consent.
* Participants must be willing to perform follow up visits for up to 5 months.
* Undergo complete blood count (CBC) with Differential and Serum Chemistry. (Results must fall within 1.5 times the normal ranges for all values for candidates to be eligible.)
* Men and Women of reproductive potential: Willingness to use approved methods of birth control or abstain from sexual intercourse from screening until removal of the AAT implants.

  * Definition of non-childbearing potential for Women: amenorrhea (previous 12 months) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
  * Definition of non-reproductive potential for Men: confirmed surgically sterile (vasectomy >3 months prior to screening).

Exclusion Criteria:

* Patients seeking elective surgery for the removal of redundant tissue from areas other than the abdomen or arm.
* Use of AAT in patients exhibiting autoimmune connective tissue disease is not recommended. When applied properly, AAT has been shown to support the migration of host cells from the surrounding tissue. Therefore, this study will exclude patients with conditions that could inhibit migration of host cells including, but not limited to, the following:

  * Fever (oral temperature >99º F at time of screening)
  * Insulin dependent diabetes
  * Low vascularity of the tissue intended for elective excision
  * Local or Systemic Infection
  * Mechanical Trauma
  * Poor nutrition or general medical condition
  * Dehiscence and/or necrosis due to poor revascularization
  * Specific or nonspecific immune response to some component of the AAT material
  * Infected or nonvascular surgical sites
  * Known cancer or receiving treatment for cancer
* Pregnant or Lactating females
* Inability to cooperate with and/or comprehend post-operative instructions
* Inability to speak or read English
* Known allergy or sensitivity to Penicillin, Streptomycin, or Amphotericin B
* Any other reason the study physicians judge would be a contraindication for receiving AAT injections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Safety of acellular adipose tissue (AAT) injections as determined by the incidence of adverse events | Up to 12 weeks post-injection
Safety of acellular adipose tissue (AAT) injections as determined by the rate of adverse events | Up to 12 weeks post-injection

SECONDARY OUTCOMES:
Assess the histopathology of explanted implants via Hematoxylin and eosin (H&E) staining | Up to 12 weeks post-injection
Assess the histopathology of explanted implants via flow cytometry | Up to 12 weeks post-injection
  Flow cytometry via fluorescence-activated cell sorting (FACS)
Assess tolerability of AAT injections per the participant-reported experience. | Up to 12 weeks post-injection
  Tolerability of AAT injections is assessed through participant-reported comfort questionnaire.

OTHER OUTCOMES:
Assess tolerability of AAT injections per the physician-reported experience. | Up to 12 weeks post-injection
  Tolerability of AAT injections is assessed through physician-reported ease-of-use with the intervention (questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer H Elisseeff, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wu I, Nahas Z, Kimmerling KA, Rosson GD, Elisseeff JH. An injectable adipose matrix for soft-tissue reconstruction. Plast Reconstr Surg. 2012 Jun;129(6):1247-1257. doi: 10.1097/PRS.0b013e31824ec3dc. PMID 22327888